CLINICAL TRIAL: NCT06523075
Title: Construction and Validation of a Sepsis Prediction Model Based on Dysregulation of Host Response
Brief Title: Host Dysregulation-Driven Sepsis Prediction Model
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: SAHoWMU-CR2024-16-214
Record Dates: First submitted 2024-07-14; First posted 2024-07-26 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis | interventions — Tumor Necrosis Factor-alpha; Interleukin-12; Interleukin-18; Complement C3; Complement C5

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sepsis Group
  Interventions: Other: Tumor Necrosis Factor; Other: Interleukin-1β; Other: Interleukin-12; Other: Interleukin-18; Other: Complement C3; Other: Complement C5
- Non-Sepsis Group
  Interventions: Other: Tumor Necrosis Factor; Other: Interleukin-1β; Other: Interleukin-12; Other: Interleukin-18; Other: Complement C3; Other: Complement C5

INTERVENTIONS:
Other: Tumor Necrosis Factor — This study is a retrospective observational study, with Tumor Necrosis Factor being one of the exposure factors under investigation.
Other: Interleukin-1β — This study is a retrospective observational study, with Interleukin-1β being one of the exposure factors under investigation.
Other: Interleukin-12 — This study is a retrospective observational study, with Interleukin-12 being one of the exposure factors under investigation.
Other: Interleukin-18 — This study is a retrospective observational study, with Interleukin-18 being one of the exposure factors under investigation.
Other: Complement C3 — This study is a retrospective observational study, with Complement C3 being one of the exposure factors under investigation.
Other: Complement C5 — This study is a retrospective observational study, with Complement C5 being one of the exposure factors under investigation.

SUMMARY:
The aim of this study is to identify risk factors associated with sepsis and to construct a predictive model for sepsis. This will provide an objective theoretical and empirical foundation for the diagnosis, assessment, and management of sepsis in our country.The primary questions addressed are:

What are the risk factors for the development of sepsis? How do we improve the prognosis of sepsis?

ELIGIBILITY:
Inclusion Criteria:

* Patients with Infection or Suspected Infection

Exclusion Criteria:

* Patients with Autoimmune Diseases
* Pregnant Women
* Patients with Advanced-Stage Cancer and Systemic Metastasis

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with Infection or Suspected Infection
Sampling Method: Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2024-10-13 (Actual); Study Completion 2024-10-17 (Actual)

PRIMARY OUTCOMES:
Sepsis | 3 months
  A rapid increase of 2 or more points points in the Sequential Organ Failure Assessment (SOFA) score after patient infection.SOFA score, which ranges from a minimum of 2 to a maximum of 15, indicates a worse outcome with higher scores.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Xiue Ye, Wenzhou, Zhejiang
  - The Second Affiliated Hospital and Yuying Children's Hospital of Wenzhou Medical University,, Wenzhou, Zhejiang